CLINICAL TRIAL: NCT02002559
Title: Endoscopic Surveillance Comparing Narrow Band Imaging (NBI) Against Lugol Chromoendoscopy for Detection of Synchronous Superficial Squamous Esophageal Neoplasia Among High Risk Patients
Brief Title: Narrow Band Imaging (NBI) Against Lugol for Squamous Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan Chiu, Professor, Chinese University of Hong Kong
Other Study IDs: 2006.077
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Superficial Esophageal Neoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NBI Magnify Endoscopy: Detection of esphageal neoplasia through recognition of brownish discolored area via NBI and characterize the lesion using IPCL upon magnifying endoscopy
- Lugol Chromoendoscopy: Detection of esophageal neoplasia through recognition of discolored area

SUMMARY:
This study aimed to compare Narrow Band Imaging (NBI) against Lugol chromoendoscopy for diagnosis of early esophageal cancers among high risk patients.

DETAILED DESCRIPTION:
The investigators recruited consecutive patients with head and neck cancers, history of squamous esophageal cancers treated by chemoradiotherapy or endoscopic resection. Endoscopic surveillance first started with NBI for detection and characterization of early esophageal cancers through observation of abnormal intrapapillary capillary loops (IPCL). Superficial esophageal neoplasia were diagnosed by IPCL Type IV, V1,V2 and Vn. Lugol chromoendoscopy would be performed subsequently and suspicious neoplasia were classified as understain or unstain lesions. The diagnostic accuracy, sensitivity and specificity of NBI were compared to Lugol chromoendoscopy with histology serving as a gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Head and Neck Cancer
2. Patients with esophageal cancer treated by chemoradiotherapy and in remission for 2 years
3. Patients with esophageal cancer treated by endoscopic resection
4. Age 18 to 80

Exclusion Criteria:

1. Allergy to Lugol iodine
2. Pregnancy
3. Previous esophagectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with Head and Neck Cancer
  2. Patients with esophageal cancer treated by chemoradiotherapy and in remission for 2 years
  3. Patients with esophageal cancer treated by endoscopic resection
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2006-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of superficial esophageal neoplasia | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Philip WY Chiu, MD, Principal Investigator — Chinese University of Hong Kong